CLINICAL TRIAL: NCT04275934
Title: Evaluation of the Impact of Self-insured Employer Implementation of an Innovative Care Model Utilizing Pharmacist-delivered MTM Services for Health Plan Beneficiaries With High Blood Pressure
Brief Title: Blood Pressure First Medication Therapy Management
Acronym: BP First
Status: Completed | Type: Observational
Sponsor: American Pharmacists Association Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 020
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypertension; Blood Pressure; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: This project will evaluate the impact of self-insured employers implementing an innovative care model utilizing pharmacist-delivered MTM services for health plan beneficiaries with high blood pressure.
  Interventions: Behavioral: Health Management; Blood Pressure

INTERVENTIONS:
Behavioral: Health Management; Blood Pressure — Pharmacists will work with the patient/study subject, referred to as the participant hereafter, and the participant's other health care providers to manage their blood pressure, making recommendations for medication and lifestyle adjustments as needed.

SUMMARY:
The primary objective of this project is to improve the health status of participants through pharmacist-delivered blood pressure control programs that demonstrate value to employers and justify adoption, sustainability and scalability of these programs.

DETAILED DESCRIPTION:
Univariate comparisons of the baseline/pre-intervention outcomes to the post-intervention outcomes will be performed on outcomes in order to determine how the intervention affects each. For continuous outcomes data the univariate comparisons of the pre-treatment and post-intervention outcomes will be performed using related samples t-test comparisons. For categorical outcomes data, comparisons of pre-intervention to post-intervention time frames will be performed using McNemar tests.

ELIGIBILITY:
Inclusion Criteria:

* All health plan beneficiaries 18 years-of-age and older
* Have filled at least one blood pressure medication in the last three months,
* Have a known hypertension diagnosis or have an uncontrolled blood pressure

Exclusion Criteria:

* Not an adult
* Not a health plan beneficiary of the self-insured employer
* Not ambulatory and able to work or participate in care visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Beneficiaries of self-insured employer who may benefit from patient-centered, team-based care that supports blood pressure control.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Control | 6-months
  Management of Systolic and Diastolic Blood Pressure Measures
Blood Pressure Change | 6-months
  Systolic and Diastolic Blood Pressure Measure Changes

SECONDARY OUTCOMES:
Blood Pressure Medication Adherence | 6-months
  Medication Adherence for Blood Pressure Medications as Measured by Proportion of Days Covered (PDC)
Health Care Utilization of Primary Care Services | 6-months
  Evaluation of Pre- and Post-Intervention Frequency of Primary Health Care Visits
Health Care Utilization of Emergency Department Services | 6-months
  Evaluation of Pre- and Post-Intervention Frequency Emergency Department Visits
Health Care Utilization of Hospital Services | 6-months
  Evaluation of Pre- and Post-Intervention Frequency of Hospital Visits

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Bluml, RPh, Principal Investigator — APhA Foundation
Locations (1):
- Woodstock Pharmaceutical & Compounding Center Inc., Woodstock, Georgia, United States